CLINICAL TRIAL: NCT04469062
Title: A Phase 3b, Randomized, Double-Blind, Parallel-Arm, Placebo- and Active- Controlled Treat-Through Study of Mirikizumab and Vedolizumab in Participants With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study of Mirikizumab (LY3074828) in Participants With Ulcerative Colitis
Acronym: LUCENT-ACT
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial was terminated secondary to a business decision, the original scientific question rendered moot by the external scientific community.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16825; I6T-MC-AMBI (Other: Eli Lilly and Company); 2019-001653-99 (EudraCT Number)
Record Dates: First submitted 2020-07-10; First posted 2020-07-13 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Ulcerative Colitis
Keywords: Interleukin-23 (IL-23) antibody; IL-23p19
MeSH Terms: conditions — Colitis, Ulcerative | interventions — mirikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mirikizumab (Experimental): Mirikizumab administered intravenously (IV) and subcutaneously (SC).
  Interventions: Drug: Mirikizumab IV; Drug: Mirikizumab SC
- Vedolizumab (Active Comparator): Vedolizumab administered IV.
  Interventions: Drug: Vedolizumab IV
- Placebo (Placebo Comparator): Placebo administered SC and IV.
  Interventions: Drug: Placebo IV; Drug: Placebo SC

INTERVENTIONS:
Drug: Mirikizumab IV — Administered IV
  Other Names: LY3074828
  Arms: Mirikizumab
Drug: Mirikizumab SC — Administered SC
  Other Names: LY3074828
  Arms: Mirikizumab
Drug: Vedolizumab IV — Administered IV
  Arms: Vedolizumab
Drug: Placebo IV — Administered IV
  Arms: Placebo
Drug: Placebo SC — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate if study drug mirikizumab is safe and effective compared to vedolizumab and placebo in participants with moderately to severely active ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of UC for at least 3 months prior to baseline
* Participants must have a confirmed diagnosis of moderately or severely active UC, as assessed by the modified Mayo score (MMS)
* Participants must have demonstrated an inadequate response to, a loss of response to, or an intolerance to conventional or to biologic therapy for UC
* Participants must, if female, meet the contraception requirements

Exclusion Criteria:

* Participants must not have a current diagnosis of Crohn's disease or inflammatory bowel disease-unclassified (indeterminate colitis)
* Participants must not have had a previous colectomy
* Participants must not have current evidence of toxic megacolon
* Participants must not have prior exposure to anti-IL-23p19 antibodies (e.g. risankizumab, brazikumab, guselkumab or tildrakizumab), vedolizumab, or natalizumab
* Participants must not have prior clinical failure or intolerance to anti-IL12p40 antibodies (e.g. ustekinumab), anti-integrin antibodies other than vedolizumab and natalizumab (e.g. etrolizumab) or anti-integrin ligand antibodies (e.g. ontamalimab) within 4 weeks prior to screening endoscopy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-20 (Estimated); Primary Completion 2024-03-13 (Estimated); Study Completion 2024-06-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants in Histologic Remission | Week 12
  Histologic remission based on histology.

SECONDARY OUTCOMES:
Percentage of Participants in Symptomatic Remission | Week 52
  Symptomatic remission based on modified Mayo Score (MMS) stool frequency (SF) and rectal bleeding (RB) subscores.
Percentage of Participants in Clinical Remission | Week 52
  Clinical remission based on MMS.
Percentage of Participants in Endoscopic Remission | Week 52
  Endoscopic remission based on MMS ES.
Percentage of Participants with Clinical Response | Week 12
  Clinical response based on MMS.
Percentage of Participants with Corticosteroid (CS) Free Remission without Surgery (Subgroup of Participants on CS at Baseline) | Week 52
  CS free remission without surgery based on clinical remission, symptomatic remission and no CS use.
Percentage of Participants with Resolution of Extraintestinal Manifestations (EIMs) Among Those That had Them at Baseline | Week 52
  Percentage of participants with resolution of EIMs among those that had them at baseline.
Change from Baseline on the Inflammatory Bowel Disease Questionnaire (IBDQ) Score | Baseline, Week 52
  Change from baseline on the IBDQ score.
Percentage of Participants Undergoing Surgery for UC (Including Colectomy) | Week 52
  Percentage of participants undergoing surgery for UC (including colectomy).
Percentage of Participants Hospitalized for UC | Week 52
  Percentage of participants hospitalized for UC.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Mirikizumab (LY3074828) in Participants With Ulcerative Colitis (LUCENT-ACT) — https://trials.lillytrialguide.com/en-US/trial/2CU7GWC1qkMxLL0Qo3HP8a